CLINICAL TRIAL: NCT02921451
Title: Prospective Analysis of Restorelle in the Treatment of Uterine Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michigan Institution of Women's Health PC (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Principal Investigator, Salil Khandwala, Medical Director, Michigan Institution of Women's Health PC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IISP 16-05
Record Dates: First submitted 2016-09-23; First posted 2016-10-03 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Uterine Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restorelle Smartmesh (Other): Surgical procedure for treatment of uterine prolapse will use the device, Restorelle Smartmesh.
  Interventions: Device: Restorelle Smartmesh

INTERVENTIONS:
Device: Restorelle Smartmesh — Patients will have surgery using the device, Restorelle Smartmesh, for treatment of uterine prolapse.

SUMMARY:
The purpose of this study is to determine the long term performance of Restorelle system for the treatment of uterine prolapse.

DETAILED DESCRIPTION:
This study is being done to evaluate the performance of the Restorelle system, which uses Smartmesh - an ultra-lightweight mesh for uterine prolapse management. Most patients undergo a hysterectomy i.e. removal of the uterus when they have a prolapse. However, this has often been found to be an unnecessary operation. The investigators are studying the use of the Restorelle mesh system to preserve the uterus when there is a uterine prolapse.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female.
2. Subject is at least 18 years of age.
3. Subjects who have already made the decision to proceed with uterine prolapse surgery using Restorelle Mesh.
4. Subject has uterine prolapse defined by Prolapse Quantification System Assessment (POPQ) score of C -2 or greater.
5. Subject reports a bothersome bulge they can see or feel per Pelvic Floor Distress Inventory Short Form 20 (PFDI-20) question 3, response of 2 or higher (i.e. response of "somewhat", "moderately" or "quite a bit").
6. Subject is willing to provide written informed consent.
7. Subject is willing and able to comply with follow-up regimen.

Exclusion Criteria:

1. Subject is pregnant or intends to become pregnant in the future.
2. Subject has a history of pelvic organ cancer (e.g. uterine, ovarian, bladder or cervical).
3. Subject has undergone any previous repair for pelvic organ prolapse.
4. Subject has undergone a hysterectomy.
5. Subject lacks competency of the English language.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients who present with recurrence of uterine prolapse following surgery as assessed by failing to meet success criteria | Within first two years after surgical procedure
  Success criteria will be defined through the examination of patient's Prolapse Quantification System Assessment (POPQ) score of C -1 or less and patient's report of bothersome bulge they can see or feel per Pelvic Floor Distress Inventory Short Form 20 (PFDI-20) question 3, response of 0 or 1 (i.e. response of "not at all"). Failure to meet this criteria will be considered recurrence of uterine prolapse.

CONTACTS AND LOCATIONS:
Overall Officials: Salil Khandwala, Principal Investigator — Advanced Urogynecology of Michigan, P.C.
Locations (1):
- Advanced Urogynecology of Michigan, P.C., Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No